CLINICAL TRIAL: NCT03451994
Title: Retrospective Analysis of Volatile Organic Compounds in Alveolar Breath as Biomarkers of Idiopathic Malodor
Brief Title: Exploratory Study of Volatile Organic Compounds in Alveolar Breath
Acronym: VOCs
Status: Completed | Type: Observational
Sponsor: Mebo Research, Inc. (Other)
Collaborators: Menssana Research, Inc. (Industry); Aurametrix (Other)
Responsible Party: Sponsor
Other Study IDs: 20111001005MEBO
Record Dates: First submitted 2018-02-18; First posted 2018-03-02 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Nutritional and Metabolic Diseases
MeSH Terms: conditions — Nutritional and Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Body odor: individuals self-reporting idiopathic body odor with or without bad breath
  Interventions: Other: Breath test
- Breath odor: individuals self-reporting idiopathic bad breath but no body odor
  Interventions: Other: Breath test

INTERVENTIONS:
Other: Breath test — Breath samples taken from all participants, analyzed with gas chromatography mass spectrometry (GC/MS), no treatment given.
  Other Names: Exhaled breath metabolomics

SUMMARY:
The purpose of this secondary analysis is to identify breath signatures associated with idiopathic malodor conditions.

DETAILED DESCRIPTION:
Individuals with metabolic disorders may sporadically produce malodors despite good hygiene. Analysis of volatile organic compounds (VOCs) helps to gain insights into medical conditions arising due to metabolic dysfunction as different metabolic pathways emit and or consume various VOCs. These VOCs can be detected via the exhaled breath collected and analyzed with a portable breath collection apparatus. VOC profiles will be compared with self-reported symptoms and other observations of participating subjects.

ELIGIBILITY:
Inclusion Criteria:

* good general health
* willing and able to travel to one of the participating sites

Exclusion Criteria:

* medical conditions that, in the opinion of the investigator, would prevent participation
* elect not to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals self-reporting idiopathic malodor production as a consequence of a systemic disorder
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2011-10-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2020-10-11 (Actual)

PRIMARY OUTCOMES:
VOCs detected | 2 years
  Expired air sample drawn principally from alveolar breath is analyzed by gas chromatography-mass spectrometry. Chromatograms are searched against the NIST library. The response for each analyte is normalized by using internal standards containing 1-bromo-4-fluoro-benzene.

SECONDARY OUTCOMES:
Correlations between breath biomarkers and self-reported observations (questionnaires) | 1 year
  VOC profiles will be compared with self-reported symptoms, observed exposures and other observations of participating subjects. Volatile organic compounds differentiating the disease activity will be identified.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Gabashvili, PhD, Principal Investigator — MeBO Research
Locations (2):
- MeBO Research, Miami, Florida, United States
- MeBO Research LTD, London, England, United Kingdom

REFERENCES:
- [Background] Phillips M. Method for the collection and assay of volatile organic compounds in breath. Anal Biochem. 1997 May 1;247(2):272-8. doi: 10.1006/abio.1997.2069. PMID 9177688